CLINICAL TRIAL: NCT05918224
Title: Streptococcus Salivarius K12 for Prevention and Treatment of Oral Mucositis in Patients Undergoing Radiotherapy for Head and Neck Tumor: A Randomized, Placebo-Controlled, Double-Blind Trial
Brief Title: Streptococcus Salivarius K12 for Prevention and Treatment of Oral Mucositis in Patients Undergoing Radiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ChiCTR2100054689
Record Dates: First submitted 2022-01-18; First posted 2023-06-26 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; nasopharyngeal carcinoma; oral mucositis; Streptococcus salivarius K12
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Carcinoma; Stomatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): S. salivarius K12 group: The S. salivarius K12 lozenges (NOW Foods, USA) contained not less than 1×109 CFU viable cells of S. salivarius K12 as the active ingredient. The S. salivarius K12 lozenges were dissolved in the mouth and then swallowed through the first day of RT to the end of treatment (1 lozenge 3 times a day).
  Interventions: Drug: Streptococcus salivarius K12
- Placebo group (Placebo Comparator): Placebo group: Placebo lozenges contained sugar and starch used as excipients in the active formulation. The placebo lozenge were dissolved in the mouth and then swallowed through the first day of RT to the end of treatment (1 lozenge 3 times a day).
  Interventions: Drug: Streptococcus salivarius K12 simulants

INTERVENTIONS:
Drug: Streptococcus salivarius K12 — The patients in intervention group were treated with Streptococcus salivarius K12 lozenges three times a day after gargling from the first day of radiotherapy up to 1 week after the end of treatment. Streptococcus salivarius K12 is dissolved in the mouth and then swallowed.
  Other Names: OralBiotic BLIS K12 (NOW Foods, USA)
  Arms: Experimental group
Drug: Streptococcus salivarius K12 simulants — Patients in control group were treated with Streptococcus salivarius K12 simulants, and its use method and use time are the same as intervention group.
  Arms: Placebo group

SUMMARY:
To evaluate the efficacy and safety of Streptococcus salivarius K12 for prevention and treatment of oral mucositis in patients undergoing radiotherapy for malignant head and neck tumors.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the efficacy and safety of Streptococcus salivarius K12 in reducing the incidence, duration, and severity of severe oral mucositis (SOM). The main questions it aims to answer are whether Streptococcus salivarius K12 can effectively prevent and treat radiation-induced oral mucositis and whether it will cause adverse events in patients undergoing radiotherapy.

Participants will be instructed to suck a Streptococcus salivarius K12 or placebo lozenge three times daily from the beginning to the end of RT. After using the lozenges, the patients should avoid eating, drinking and conducting any oral hygiene activities for at least 1 hour.

Researchers will compare Streptococcus salivarius K12 group and placebo group to see if oral probiotic are beneficial in preventing and treating oral mucositis in patients undergoing radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-metastatic head and neck malignant tumor diagnosed by histopathology;
* Aged 18 to 80 years;
* Systemic functional status Eastern Cooperative Oncology Group (ECOG) (Appendix 1) rating ≤2;
* Receiving definitive RT or postoperative adjuvant RT at a dose of 60-72Gy with/without concurrent chemotherapy;
* Sign the informed consent

Exclusion Criteria:

* Patients with known allergy to probiotic or severe allergic constitution;
* Using antibiotics/antifungal drugs within 1 month or using antimicrobial mouthwash within 1 week before the study;
* Poor oral hygiene and/or severe periodontal diseases;
* Any previous RT to the head and neck region;
* Deemed unsuitable for the study by the investigators (concomitant with any other severe diseases).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The incidence of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  Oral mucositis is assessed by trained physicians according to World Health Organization (WHO) oral toxicity Scale.

SECONDARY OUTCOMES:
Taste function | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks); and 1, 3, 6, 9 and 12 months after the end of radiotherapy
  Electrogustometer test and taste strips test.
Xerostomia | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks); and 1, 3, 6, 9 and 12 months after the end of radiotherapy
  Patients self-rated xerostomia according to summated xerostomia inventory (SXI), and researchers measured saliva flow rates.
functional assessment of cancer therapy-head and neck (FACT- H&N) quality of life questionnaire. | 1 week before radiotherapy; at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks); ; and 1, 3, 6, 9 and 12 months after the end of radiotherapy
  FACT- H&N quality of life questionnaire.
Adverse events | From the first day of radiotherapy to the day of the last radiation dose received, usually 6 or 6.5 weeks
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version
The duration of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  The first determination of SOM to the first instance of non-severe OM (WHO grade <3), without a subsequent instance of SOM. Patients without observed SOM were assigned a duration of 0 days.
The time to onset of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  Time from the first day of radiotherapy to the first determination of SOM. Patients without observed SOM were assigned onset days of 6 or 6.5 weeks.
The number of patients who missed five or more consecutive radiation fractions. | The time period is the period from the start of radiotherapy to the completion of radiotherapy
  The number of patients who missed five or more consecutive radiations and the reasons for this are recorded during radiotherapy.
Mouth and throat soreness (MTS) scores | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6 1/2 weeks
  Patients report mouth and throat soreness (MTS) scores (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms.
Oral activities scores | The time period is the period from the start of radiotherapy to the completion of radiotherapy. The evaluation period is approximately 6 weeks and 6 1/2 weeks
  Patients report the degree to the impact of MTS on oral activities (including swallowing, drinking, eating, talking, sleeping) (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No